CLINICAL TRIAL: NCT05003791
Title: Perceived Social Support, Heart Rate Variability, and Hopelessness in Patients With Ischemic Heart Disease
Acronym: Hope Beats
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Sigma Theta Tau International (Other)
Responsible Party: Principal Investigator, Madison (Buursma) Goodyke, Principal Investigator, University of Illinois at Chicago
Other Study IDs: 2021-0544; F31NR019714 (NIH)
Record Dates: First submitted 2021-07-12; First posted 2021-08-12 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Heart Disease
Keywords: heart rate variability; hopelessness; perceived social support
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease is the leading cause of death worldwide, with ischemic heart disease (IHD) the leading cause of cardiovascular mortality. Persons with IHD suffering from psychological distress, including hopelessness, are more likely to die from IHD. Following a stressful event, the vagus nerve enables activation of either a sympathetic (fight/flight) or parasympathetic (rest/digest) response. Heart rate variability (HRV), the beat-to-beat variability between normal successive heart beats, is a biomarker of both adaptive and maladaptive reactions to stress. Decreased HRV predicts greater risk for morbidity and mortality and is associated with poor mental health outcomes in persons with IHD. As stated by polyvagal theory, HRV may be influenced by social support. Decreased perceived social support (PSS), a social determinant of cardiovascular risk, is predictive of increased morbidity and mortality in persons with IHD. Decreased PSS has been associated with hopelessness in patients with cancer, but this relationship has not been studied in IHD beyond the applicant's small pilot study of patients with hopelessness. Hopelessness, a negative outlook and sense of helplessness about the future, is present in 27-52% of patients with IHD. This is of grave concern, because hopelessness is associated with a 3.4 times increased risk of mortality and nonfatal myocardial infarction in patients with IHD, independent of depression. This research focuses on understanding the biological (HRV) and social (PSS) aspects of hopelessness, with the long-term goal of developing and testing novel interventions to reduce the adverse effects of hopelessness and improve health outcomes in patients with IHD. Participants for this cross-sectional study will be recruited while hospitalized for an IHD event. Participants will include patients who report moderate to severe hopelessness from the sponsor's NIH-funded study (n = 225); additional patients with minimal to no hopelessness will be recruited and enrolled by the applicant (n = 45). Data collection will take place remotely two weeks after hospital discharge. Specific aims include: Aim 1) Evaluate the relationship between HRV and hopelessness in patients with IHD; Aim 2) Determine the relationship between PSS and hopelessness in patients with IHD; and Aim 3) Explore the possible mediating effect of HRV on the relationship between PSS and hopelessness in patients with IHD.

DETAILED DESCRIPTION:
Design, Sample, and Setting. A cross-sectional design will be used to address study aims. Data will be collected 2 weeks after hospital discharge for an IHD event. Patients who provide written-informed consent and enroll will be sent a package with study materials to their home and complete a phone visit 2 weeks after hospital discharge. Comorbidities and clinical characteristics will be abstracted from the medical record. Recruitment and enrollment of all patients will take place during patients' hospitalization for an IHD event at a large teaching hospital in the Midwestern United States. The applicant will analyze data from Dr. Dunn's NIH-funded study (R01NR017649) of 225 patients with IHD who report moderate to severe hopelessness and will additionally recruit 45 sex and age matched patients with IHD who report minimal to no hopelessness.

Recruitment, Screening and Consent. Study enrollers, employed by the recruiting hospital, will determine eligibility for hopelessness screening by reviewing the patient's medical record. Eligible hospitalized IHD patients will be called by enrollers and invited to screen for hopelessness over the phone. Enrollers will use a script to introduce the screening portion of the study, explaining that eligibility for Dr. Dunn's study (enrolling those who report moderate to severe hopelessness) and the applicant's study (enrolling those with minimal or no hopelessness) will depend on screening results. Interested patients will provide consent for the hopelessness screening, including a HIPAA waiver. Patients who provide consent will be screened for hopelessness using the 10-item state subscale of the 23-item State-Trait Hopelessness Scale (STHS). Based on published cut-point criteria, a criterion of ≥ 1.8 will be used for classification of moderate to severe hopelessness levels. Patients who score ≥ 1.8 during screening will be asked to participate in Dr. Dunn's study, and the applicant will have access to this data. Patients who score < 1.8 on the STHS will be asked by the applicant to participate in the proposed research. To mitigate potential exposure to COVID-19, the only in-person contact with participants throughout the course of the proposed study will be during the enrollment process. During enrollment, the applicant will explain the study, risks, benefits, voluntary nature of participation, and the patient's right to discontinue participation at any time without consequences. Written consent will be obtained.

Data Collection Procedures. Study participants will receive the study package by USPS mail two weeks after hospital discharge and will also receive a phone visit at Week 2. Study package materials will include a Polar H7 heart rate monitor, ActiGraph wGT3X-BT (to link to the Polar monitor for HRV data collection), written instructions for HRV measurement, hard copies of questionnaires (to view during the data collection phone call), instructions to return the monitors, and a prepaid return envelope. Participants will also be sent a secure link via text or email to an instructional video depicting verbal and visual demonstration of proper HRV measurement. The applicant will call the participant once a mail delivery notice has been received to instruct and confirm proper placement of the monitors used to measure HRV and answer any questions. All data collection will occur at Week 2.

HRV Procedures. At Week 2, participants will be instructed to place the Polar H7 heart rate monitor around the center of their chest, in contact with the skin, and the ActiGraph wGT3X-BT around their waist, according to directions outlined in the written instructions provided and as demonstrated in the instructional video and practiced with the applicant over the phone. Participants will be informed that the monitors are used to gather data about their body at rest. The Polar H7 heart rate monitor connects to the ActiGraph with Bluetooth® wireless technology so that the interval between normal to normal (RR) heart beats can be transferred to csv files for analysis. The Polar H7 has demonstrated strong correlation with ECG for measuring HRV (r=0.99). The HRV protocol will take place during a 10-minute time period on two consecutive days, to ensure at least one timeframe of usable data. Participants will be instructed to place the monitors first thing in the morning after they wake up and empty their bladder. Once the monitors are placed, participants will be instructed to lay supine, still, and quiet for 10 minutes. The standardized HRV protocol enhances reliability of the HRV measurement because control of extraneous variables is maintained. Respirations will not be controlled because this can artificially increase HF HRV. The gold standard amount of time for a short-term HRV recording is 5 minutes. The intermediate 5 minutes of the recording will be used for analysis, so that the initial minutes of lying flat and the final minutes will be removed. After the participant completes the two HRV measurements, they will be asked to return the monitors in a prepaid envelope that will be picked up from their mailbox by USPS, mitigating any exposure to COVID-19.

Phone Visit to Complete Questionnaires. After completion of the HRV measurement instructional phone visit, participants will receive their Week 2 data collection visit. Participants in Dr. Dunn's study will receive their phone visit from a trained data collector prior to the RCT's intervention. Participants in the applicant's study will receive their phone visit from the applicant. The data collectors/applicant will follow identical scripts for data collection. During the phone visit, the data collector/applicant will first ask how HRV measurement went that morning and remind participants to complete the measurement the following morning. Participants will then complete four questionnaires. Deidentified HRV data will be uploaded into Box, a secure cloud-based storage service, by the applicant. All questionnaire and electronic medical record data will be logged directly into REDCap using a secure electronic tablet.

Measures. The following questionnaires will be completed during the data collection phone visit. Demographic Questionnaire: Demographics are being collected to describe the sample and determine if these variables are confounders. State-Trait Hopelessness Scale (STHS): The STHS measures state and trait hopelessness. The scale uses a 4-point Likert-type scale ranging from 1 (strongly disagree) to 4 (strongly agree). Item scores are added and divided by the number of items to provide a total score for each subscale, ranging in a final score from 1-4 with higher scores indicating greater levels of hopelessness. In patients with IHD, the scale has demonstrated reliability and validity. ENRICHD Social Support Inventory (ESSI): The ESSI measures PSS. The ESSI is a 7-item instrument that uses a 5-point Likert-type scale for items 1-6 ranging from 1 (none of the time) to 5 (all of the time). The 7th item is yes/no. Items are summed for a final score with a range from 8-34, higher scores indicate greater levels of PSS. The ESSI was found to be valid and reliable in patients with IHD. Patient Health Questionnaire 9 (PHQ-9): The PHQ-9 measures depressive symptom severity. The instrument is comprised of 9 items that are scored on a Likert-type scale ranging from 0 (not at all) to 3 (nearly every day). Item scores are summed for a total score ranging from 0-27, higher scores indicating greater depressive symptom severity. The PHQ-9 has been validated in patients with IHD. Internal reliability and criterion and construct validity have been previously established. Depressive symptoms are being measured as a potential covariate because of the known association between hopelessness and depression.

Both a medical record abstraction and the Charlson Comorbidity Index are completed within two weeks after the participant's hospital discharge. The medical record abstraction is completed to obtain participant clinical characteristics. The Charlson Comorbidity Index is a prognostic index of comorbidity. The instrument predicts 1-year mortality based on illness severity, reason for admission, and weighted comorbidity score. It is a reliable and valid prognostic indicator for in-hospital and 1-year outcomes in patients with IHD.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old; diagnosed with myocardial infarction, unstable angina, or undergoing percutaneous coronary intervention or coronary artery bypass graft surgery; and speak and read English.

Exclusion Criteria:

* The following exclusion criteria are in place for Aims 1 and 3 because they affect HRV: having a pacemaker or implanted cardioverter-defibrillator, chronic arrhythmia, history of or current valvular disease, history of organ transplant, current use of immunosuppressive medications, or diabetic autonomic insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected 2 weeks after hospital discharge for an IHD event. Patients who provide written-informed consent and enroll will be sent a package with study materials to their home and complete a phone visit 2 weeks after hospital discharge. Recruitment and enrollment of all patients will take place during patients' hospitalization for an IHD event at a large teaching hospital in the Midwestern United States.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madison Goodyke, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
All informed consent documents will include a statement informing participants that the study will be registered at ClinicalTrials.gov. Data sets and associated documentation including protocols, procedures, and instruments will be provided. The data sets will include all data collected at the Week 2 visit and chart review. Data will only be made available under terms and conditions consistent with the informed consent provided by the individual participants, and as approved by the University of Illinois at Chicago IRB and any local, state, and federal laws and regulations. To reduce the likelihood that any individual participant can be identified and to safeguard privacy, all personal identifiers will be deleted from all data sets. Original ID numbers will be replaced with new, randomized ID numbers to sever linkage with existing data both in terms of the ID number and order within the data. The data set will be prepared in accordance with guidelines for the data repository.

REFERENCES:
- [Derived] Goodyke MP, Tintle N, Collins E, DeVon HA, Bronas UG, Baynard T, Dunn SL. Lower Perceived Social Support Associated With Greater Hopelessness in Patients After an Acute Ischemic Heart Disease Event. J Cardiovasc Nurs. 2025 Sep-Oct 01;40(5):E239-E247. doi: 10.1097/JCN.0000000000001163. Epub 2024 Oct 24. PMID 39454079
- [Derived] Goodyke MP, Bronas UG, Baynard T, Tintle N, DeVon HA, Collins E, Dunn SL. Relationships Among Heart Rate Variability, Perceived Social Support, and Hopelessness in Adults With Ischemic Heart Disease. J Am Heart Assoc. 2024 Feb 20;13(4):e032759. doi: 10.1161/JAHA.123.032759. Epub 2024 Feb 13. PMID 38348815

RESULTS

PARTICIPANT FLOW:
Groups:
- Hope Beats: Participants that met the inclusion criteria and screened as experiencing none to mild hopelessness (a score of < 1.8 on the State-Trait Hopelessness Scale) and were enrolled in the Hope Beats study
Period: Overall Study
Arm/Group | Hope Beats
Started | 48
Completed | 45
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Hope Beats
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.44 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45
State Hopelessness Screening [Mean (Standard Deviation); unit: units on a scale] — Participants state hopelessness score on the State Trait Hopelessness Scale (STHS) during study screening. The STHS uses a Likert-type scale ranging from 1 (strongly disagree) to 4 (strongly agree) and differentiates state and trait hopelessness. For the 10-item state subscale, participants respond to statements based on how they feel "today (right now)." The responses for each subscale are totaled and divided by the number of items in the subscale to provide a final score ranging from one to four, with lower scores indicating lower levels of hopelessness.
  units on a scale | 1.25 (0.21)
Trait Hopelessness [Mean (Standard Deviation); unit: units on a scale] — Participants trait hopelessness score on the State Trait Hopelessness Scale (STHS) during study screening. The STHS uses a Likert-type scale ranging from 1 (strongly disagree) to 4 (strongly agree) and differentiates state and trait hopelessness. For the 13-item trait subscale, responses are based on how participants feel "typically (over the years)." The responses for each subscale are totaled and divided by the number of items in the subscale to provide a final score ranging from one to four, with lower scores indicating lower levels of hopelessness.
  units on a scale | 1.41 (0.36)
Perceived Social Support [Mean (Standard Deviation); unit: units on a scale] — Using the 5-item ENRICHD Social Support Inventory (ESSI). The ESSI uses a Likert-type scale ranging from 1 (none of the time) to 5 (all of the time). Responses for each item are summed for a final score ranging from 5-25 for the 5-item version. Higher scores indicate greater levels of perceived social support.
  units on a scale | 23.16 (2.92)
Depressive Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Measured using the Patient-Health Questionnaire-9 (PHQ-9). Items on the PHQ-9 are scored on a Likert-type scale from 0 (not at all) to 3 (nearly every day). Responses are summed for a total score ranging from 0-27, with lower scores indicating less depressive symptom severity.
  units on a scale | 4.09 (3.84)
High frequency heart rate variability [Mean (Standard Deviation); unit: log(ms^2)] — Log transformed short-term (5 minute) measurement of HF HRV Population: Analyzed all participants with appropriate HRV data. These are all the participants with an HRV recording of at least 5 minutes in length with less than 5% artifact corrected.
  log(ms^2)
    number analyzed (Participants) | 37
    (all) | 4.15 (1.19)
RMSSD heart rate variability [Mean (Standard Deviation); unit: log(ms)] — Log transformed short-term (5 minute) measurement of RMSSD HRV Population: Analyzed all participants with appropriate HRV data. These are all the participants with an HRV recording of at least 5 minutes in length with less than 5% artifact corrected.
  log(ms)
    number analyzed (Participants) | 37
    (all) | 2.72 (0.63)
History of depression [Count of Participants; unit: Participants] | 13
Has insurance [Count of Participants; unit: Participants] | 41
Married [Count of Participants; unit: Participants] | 36
Employed [Count of Participants; unit: Participants] | 26
Completed some college or more schooling [Count of Participants; unit: Participants] | 41
Had coronary artery bypass graft surgery during hospitalization [Count of Participants; unit: Participants] | 24
Prescribed a beta-blocker at time of discharge [Count of Participants; unit: Participants] — Population: Only documented beta-blocker prescription for participants with useable HRV data.
  Participants
    number analyzed (Participants) | 37
    (all) | 31

OUTCOME MEASURES:

1. Primary Outcome: State Hopelessness
Description: The State-Trait Hopelessness Scale (STHS) was used to measure state hopelessness. The STHS uses a Likert-type scale ranging from 1 (strongly disagree) to 4 (strongly agree) and differentiates state and trait hopelessness. For the 10-item state subscale, participants respond to statements based on how they feel "today (right now)." The responses for each subscale are totaled and divided by the number of items in the subscale to provide a final score ranging from one to four, with lower scores indicating lower levels of hopelessness.
Time Frame: baseline data was obtained two weeks after hospital discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hope Beats
Number analyzed (Participants) | 45
units on a scale | 1.25 (0.21)
Statistical Analysis 1: Comparison: Hope Beats; Test type: Other — This was a cross-sectional design; p < 0.05, Regression, Linear

2. Primary Outcome: Log Transformed High Frequency Heart Rate Variability
Description: Participants completed a short-term heart rate variability (HRV) measurement at rest while laying supine, silent, and still for 10 minutes. From the 10-minute HRV recordings, the 5-minute intermediate segment with the least amount of artifact was used for analysis. Kubios HRV Software was used to analyze the HRV data. Kubios utilizes Fast Fourier Transform to run frequency domain analyses. Artifact were identified and corrected using a threshold-based artifact correction algorithm in Kubios that compares RR intervals against a local average interval. The lowest level threshold thought to detect artifact without overcorrecting normal beats was utilized for each recording. Only recordings with < 5% artifact were used in the analysis
Time Frame: Baseline data was obtained 2 weeks after hospital discharge
Population: All participants with a useable 5 minute short-term HRV recording with less than 5% corrected artifact
Measure: Mean (Standard Deviation); unit: log(ms^2)
Arm/Group | Hope Beats
Number analyzed (Participants) | 37
log(ms^2) | 4.15 (1.19)
Statistical Analysis 1: Comparison: Hope Beats; Test type: Other — This was a cross-sectional design; p < 0.05, Regression, Linear

3. Primary Outcome: Log Transformed Root Mean Square of Successive Differences Between Normal Heartbeats
Description: Participants completed a short-term heart rate variability (HRV) measurement at rest while laying supine, silent, and still for 10 minutes. From the 10-minute HRV recordings, the 5-minute intermediate segment with the least amount of artifact was used for analysis. Kubios HRV Software was used to analyze the HRV data. Artifact were identified and corrected using a threshold-based artifact correction algorithm in Kubios that compares RR intervals against a local average interval. The lowest level threshold thought to detect artifact without overcorrecting normal beats was utilized for each recording. Only recordings with < 5% artifact were used in the analysis
Time Frame: Baseline data was obtained 2 weeks after hospital discharge
Population: All participants with a useable 5 minute short-term HRV recording with less than 5% corrected artifact.
Measure: Mean (Standard Deviation); unit: log(ms)
Arm/Group | Hope Beats
Number analyzed (Participants) | 37
log(ms) | 2.72 (0.63)
Statistical Analysis 1: Comparison: Hope Beats; Test type: Other — This was a cross-sectional design; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Hope Beats
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT05003791/Prot_SAP_000.pdf